CLINICAL TRIAL: NCT05823389
Title: The Use of Flapless Enamel Matrix Derivative in Treating Periodontal Residual Pockets: A Single-centre Randomized Clinical Trial
Brief Title: Flapless Emdogain in the Treatment of Periodontal Residual Pockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Mahmoud Abu-Ta'a, Associate Professor, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMD
Record Dates: First submitted 2023-04-07; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Chronic Periodontitis, Generalized
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flapless Emdogain (FEMD) group (Experimental): Re-instrumentation with flapless emdogain application
  Interventions: Procedure: Re-instrumentation with flapless Emdogain application
- Placebo group (Active Comparator): Re-instrumentation without flapless emdogain application
  Interventions: Procedure: Re-instrumentation with placebo application

INTERVENTIONS:
Procedure: Re-instrumentation with flapless Emdogain application — Teeth with deep probing pocket depths were randomized to receive re-instrumentation with adjunctive flapless administration of EMD
  Arms: Flapless Emdogain (FEMD) group
Procedure: Re-instrumentation with placebo application — Teeth with deep probing pocket depths were randomized to receive re-instrumentation with adjunctive placebo application
  Arms: Placebo group

SUMMARY:
48 adult patients participated in a single-centre randomized clinical trial with split- mouth design. They had presented at re-evaluation after initial non-surgical periodontal therapy (steps 1 and 2 of periodontal therapy) for generalized periodontitis with at least 2 teeth with residual probing pocket depths (PPD) ≥5 and ≤8 mm, with bleeding on probing (BOP). Two teeth with similar PPD were randomized to receive re-instrumentation either with (test) or without (control) adjunctive flapless administration of EMD. Differences in the changes of PPD and BOP from baseline to 6 and 12 months will be analysed, and the frequencies of pocket closure (PPD ≤4 mm and no BOP) will be compared

ELIGIBILITY:
Inclusion Criteria:

* at least two residual pockets with probing pocket depth (PPD) ≥5 and ≤8 mm,
* bleeding on probing (BOP),
* mobility ≤degree 1 and
* no furcation involvement.

Exclusion Criteria:

* full mouth plaque score >20%,
* uncontrolled systemic disease,
* history of malignant disease in the oral cavity or previous radiotherapy in the head or neck area,
* pregnant or lactating females,
* drug and alcohol abuse,
* smoking >10 cigarettes per day and
* inadequate restorative therapy or malocclusion.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Differences in changes of probing pocket depths (PPD) from baseline to 6 and 12 months | 12 months
  probing pocket depth (PPD)
Differences in changes of bleeding on probing (BOP) from baseline to 6 and 12 months | 12 months
  bleeding on probing (BOP)

SECONDARY OUTCOMES:
frequencies of pocket closure | 12 months
  PPD ≤4 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Arab American University, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided